CLINICAL TRIAL: NCT02043847
Title: BMT-03: A Phase I Trial of Total Marrow Irradiation in Addition to High Dose Melphalan Conditioning Prior to Autologous Transplant for Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: TMI With HD Mel in ASCT for R/R Multiple Myeloma (BMT-03)
Acronym: BMT-03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Damiano Rondelli, MD, Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0201; 2013-0201 (Other: UIC Office for the Protection of Research Subjects (OPRS))
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2024-10-21 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma, Relapsed; Multiple Myeloma, Refractory to Standard Treatment
Keywords: Multiple Myeloma; Relapsed; Refractory; Progressive Disease; Symptomatic
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Disease Progression | interventions — Melphalan; Filgrastim; Granulocyte Colony-Stimulating Factor; Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: Increasing doses of Total Marrow Irradiation (TMI), 3 Gy, 6 Gy, and 9 Gy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1Total Marrow Irradiation (TMI) 3Gy (Experimental): 3Gy with standard high dose melphalan prior to autologous stem cell rescue
  Interventions: Radiation: Total Marrow Irradiation; Drug: Melphalan; Drug: Filgrastim (G-CSF); Procedure: Autologous transplant
- Cohort 2 Total Marrow Irradiation (TMI) 6Gy (Experimental): 6Gy with standard high dose melphalan prior to autologous stem cell rescue
  Interventions: Radiation: Total Marrow Irradiation; Drug: Melphalan; Drug: Filgrastim (G-CSF); Procedure: Autologous transplant
- Cohort 3 Total Marrow Irradiation (TMI) 9Gy (Experimental): 9Gy with standard high dose melphalan prior to autologous stem cell rescue
  Interventions: Radiation: Total Marrow Irradiation; Drug: Melphalan; Drug: Filgrastim (G-CSF); Procedure: Autologous transplant

INTERVENTIONS:
Radiation: Total Marrow Irradiation — Subjects in this trial will receive total marrow irradiation 3Gy per day for up to four days and as little as one day
  Arms: Cohort 1Total Marrow Irradiation (TMI) 3Gy
Drug: Melphalan — Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning therapy prior to transplant
  Other Names: Alkeran ®
  Arms: Cohort 1Total Marrow Irradiation (TMI) 3Gy
Drug: Filgrastim (G-CSF) — Subjects to begin GCSF 5 μg/kg/d SC or IV on Day 5 and continue until ANC > 1000/mm^3 over period of 3 days.
  Other Names: Neupogen®
  Arms: Cohort 1Total Marrow Irradiation (TMI) 3Gy
Procedure: Autologous transplant — Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning with autologous stem cell rescue
  Arms: Cohort 1Total Marrow Irradiation (TMI) 3Gy
Radiation: Total Marrow Irradiation — Subjects in this trial will receive total marrow irradiation 6Gy per day for up to four days and as little as one day
  Arms: Cohort 2 Total Marrow Irradiation (TMI) 6Gy
Drug: Melphalan — Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning therapy prior to transplant
  Other Names: Alkeran ®
  Arms: Cohort 2 Total Marrow Irradiation (TMI) 6Gy
Drug: Filgrastim (G-CSF) — Subjects to begin GCSF 5 μg/kg/d SC or IV on Day 5 and continue until ANC > 1000/mm^3 over period of 3 days
  Other Names: Neupogen®
  Arms: Cohort 2 Total Marrow Irradiation (TMI) 6Gy
Procedure: Autologous transplant — Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning with autologous stem cell rescue
  Arms: Cohort 2 Total Marrow Irradiation (TMI) 6Gy
Radiation: Total Marrow Irradiation — Subjects in this trial will receive total marrow irradiation 9Gy per day for up to four days and as little as one day
  Arms: Cohort 3 Total Marrow Irradiation (TMI) 9Gy
Drug: Melphalan — Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning therapy prior to transplant
  Other Names: Alkeran ®
  Arms: Cohort 3 Total Marrow Irradiation (TMI) 9Gy
Drug: Filgrastim (G-CSF) — Subjects to begin GCSF 5 μg/kg/d SC or IV on Day 5 and continue until ANC > 1000/mm^3 over period of 3 days
  Other Names: Neupogen®
  Arms: Cohort 3 Total Marrow Irradiation (TMI) 9Gy
Procedure: Autologous transplant — Subjects will receive standard melphalan 200mg/m^2 (100mg/m^2 day-2 and day-1) conditioning with autologous stem cell rescue
  Arms: Cohort 3 Total Marrow Irradiation (TMI) 9Gy

SUMMARY:
In this phase I trial, patients with relapsed or refractory multiple myeloma will receive standard autologous stem cell transplant conditioned with high dose melphalan. In addition to Melphalan, the conditioning will include targeted total marrow irradiation (TMI). This is a conventional 3+3 phase I trial with increasing doses of TMI from minimum 3Gy to Maximum 9Gy.

DETAILED DESCRIPTION:
In this phase I trial, patients with relapsed or refractory multiple myeloma will receive standard high dose melphalan with autologous stem cell rescue. In addition the pre-transplant conditioning will include targeted total marrow irradiation (TMI). This conventional 3+3 phase I trial will increase the dose of TMI until the maximum tolerated dose (MTD) is reached. Initial patients enrolled will receive the lowest possible dose of 3Gy. Maximum dose will be 9Gy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting criteria for symptomatic myeloma
2. Patients who have progressive myeloma following initial induction (patients may have received any number of treatment regimens including prior autologous transplant)
3. Patient age 18-75 years at time of enrollment
4. Karnofsky performance status of ≥70
5. Cardiac function: LVEF >40%
6. Hepatic: Bilirubin <2x upper limit of normal and ALT and AST < 2.5x the upper limit of normal
7. Renal: Creatinine clearance of >30mL/min, estimated or calculated
8. Pulmonary: DLCO, FEV1, FVC >50% of predicted (after correction for hemoglobin)

Exclusion Criteria:

1. Patients with diagnosis of plasma cell leukemia
2. Patients with truly non secretory myeloma (patients with light chain disease are eligible)
3. Pregnant or breast-feeding
4. Uncontrolled viral, fungal or bacterial infection Note: Infection is permitted if there is evidence of response to medication. Eligibility of HIV infected patients will be determined on a case-by-case basis.
5. Patients who have undergone prior allogeneic stem cell transplant
6. Prior solid organ transplant
7. Patients receiving prior radiation to more than 20% of bone marrow containing areas

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Rondelli, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Patel P, Oh AL, Koshy M, Sweiss K, Saraf SL, Quigley JG, Khan I, Mahmud N, Hacker E, Ozer H, Peace DJ, Weichselbaum RR, Aydogan B, Rondelli D. A phase 1 trial of autologous stem cell transplantation conditioned with melphalan 200 mg/m2 and total marrow irradiation (TMI) in patients with relapsed/refractory multiple myeloma. Leuk Lymphoma. 2018 Jul;59(7):1666-1671. doi: 10.1080/10428194.2017.1390231. Epub 2017 Oct 25. PMID 29065747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1Total Marrow Irradiation (TMI) 3Gy | Cohort 2 Total Marrow Irradiation (TMI) 6Gy | Cohort 3 Total Marrow Irradiation (TMI) 9Gy
Started | 3 | 3 | 6
Completed | 1 | 0 | 0
Not Completed | 2 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1Total Marrow Irradiation (TMI) 3Gy | Cohort 2 Total Marrow Irradiation (TMI) 6Gy | Cohort 3 Total Marrow Irradiation (TMI) 9Gy | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 4 | 6
  >=65 years | 1 | 3 | 2 | 6
Age, Continuous [Mean (Full Range); unit: Years] | 59 [56 to 66] | 68 [66 to 69] | 58 [40 to 71] | 61 [40 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4
  Male | 3 | 1 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 1 | 1 | 5 | 7
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 1 | 1 | 4 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Gy
Description: Assessing MTD of TMI of 3Gy, 6Gy and 9Gy
Time Frame: Up to 60 days post-transplant.
Population: 3 participants received 3Gy, 3 participants received 6Gy and 6 participants received 9Gy
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 12
Participants | NA — To clarify there was an insufficient number of events to determine the MTD

2. Secondary Outcome: Progression Free Survival (PFS) and in Patients With Multiple Myeloma (Relapsed or Refractory) Undergoing Autologous Stem Cell Transplant Using the Combination of High Dose Melphalan and Total Marrow Irradiation
Description: The disease status of enrolled patients will be evaluated based on the International Myeloma Working Group Criteria.
  Response Criteria
  Stringent Complete Response (sCR) in addition to CR all of the following:
  1. Normal free light chain ratio (FLC)
  2. Absence of clonal cells in the bone marrow by immunohistochemistry if this is performed
  Complete Response (CR) requires all of the following:
  1. Absence of the original monoclonal paraprotein in the serum or the urine by routine electrophoresis and by immunofixation. The presence of new monoclonal bands consistent with oligoclonal immune reconstitution does not exclude CR.
  2. Less than 5% plasma cells in a bone marrow aspirate and bone marrow biopsy if this is performed.
  3. No increase in size or number of lytic bone lesions on radiologic investigation (development of compression fracture does not exclude CR and radiographs are not required to document CR if not clinically indicated)
  4. Disappearance of soft tissue plasmacytoma
Time Frame: Up to 1 year post-transplant.
Population: There was no MTD reached for any Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1Total Marrow Irradiation (TMI) 3Gy | Cohort 2 Total Marrow Irradiation (TMI) 6Gy | Cohort 3 Total Marrow Irradiation (TMI) 9Gy
Number analyzed (Participants) | 3 | 3 | 6
Participants | 1 | 1 | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cohort 1Total Marrow Irradiation (TMI) 3Gy | Cohort 2 Total Marrow Irradiation (TMI) 6Gy | Cohort 3 Total Marrow Irradiation (TMI) 9Gy
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/6
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1Total Marrow Irradiation (TMI) 3Gy (N=3) | Cohort 2 Total Marrow Irradiation (TMI) 6Gy (N=3) | Cohort 3 Total Marrow Irradiation (TMI) 9Gy (N=6)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) — Metastatic prostate cancer(3GY) Progressive myeloma (6Gy and 9Gy)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1Total Marrow Irradiation (TMI) 3Gy (N=3) | Cohort 2 Total Marrow Irradiation (TMI) 6Gy (N=3) | Cohort 3 Total Marrow Irradiation (TMI) 9Gy (N=6)
Mucositis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No